CLINICAL TRIAL: NCT03507465
Title: Letrozole Plus Low-Dose Metronomic Capecitabine Versus EC-T (Epirubicin/Cyclophosphamide Followed by Docetaxel) as Neoadjuvant Therapy for ER+/HER2-negative Breast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Guangdong General Hospital
Record Dates: First submitted 2018-04-15; First posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: letrozole; metronomic; capecitabine; neoadjuvant; chemotherapy; ER+/HER2-
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letrozole Plus Low-Dose Metronomic Capecitabine (Experimental)
  Interventions: Drug: Letrozole Plus Low-Dose Metronomic Capecitabine
- EC-T (Active Comparator)
  Interventions: Drug: EC-T

INTERVENTIONS:
Drug: Letrozole Plus Low-Dose Metronomic Capecitabine — Letrozole Plus Low-Dose Metronomic Capecitabine
  Arms: Letrozole Plus Low-Dose Metronomic Capecitabine
Drug: EC-T — Epirubicin/Cyclophosphamide Followed by Docetaxel
  Arms: EC-T

SUMMARY:
Patients with ER+/HER2- breast cancer (presumably the luminal A subtype) could potentially avoid the standard chemotherapy use. Letrozole Plus Low-Dose Metronomic Capecitabine may offer similar efficacy and less toxicity to standard chemotherapy in ER+/HER2- breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

-women (age 18-70 years) with clinical T2-3 N0-1 M0 ER-positive (ER) allred score 4-8，and progesterone receptor-positive (PgR) ，HER2-negative adequate bone marrow reserve (WBC count, 3.5 *109/L; platelets, 100*109/L; hemoglobin, 10g/dL), hepatic function (AST/ALT bilirubin and alkaline phosphatase levels 1.25 the upper limit of normal value), and renal function (serum creatinine 1.25 the upper limit of normal value).

Luminal A/ lymph node positive breast cancer or Luminal B breast cancer patients

Exclusion Criteria:

* (a) male patients; (b) patients with inflammatory breast cancer or distant metastasis; (c) patients who were previously treated with chemotherapy, radiation therapy or prior treatment with AIs or antiestrogens for breast cancer; (d) patients with a second concomitant neoplasm; and (e) patients who could not meet the eligibility criteria.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-11-29 (Estimated); Study Completion 2020-11-29 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 6 month
  objective response rate (ORR) measured by breast ultrasound monthly

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li WP, Zhu T, Hu MX, Yang M, Ji F, Gao HF, Yang CQ, Zhang LL, Cheng MY, Xu FP, Wang K. Comparison of the efficacy and safety of the EC-T (epirubicin/cyclophosphamide followed by docetaxel) and TCb (docetaxel/carboplatin) neoadjuvant regimens in early TOP2A-normal stage II-III breast cancer. Neoplasma. 2020 Nov;67(6):1409-1415. doi: 10.4149/neo_2020_200130N96. Epub 2020 Jul 13. PMID 32657611